CLINICAL TRIAL: NCT06030895
Title: Pharmacogenetic Study of Sorafenib In Egyptian Patients With Hepatocellular Carcinoma.
Brief Title: Sorafenib In Egyptian Patients With Hepatocellular Carcinoma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sorafenib In Egyptian Patients
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: ATG10; IL6; Genotyping; Safety; Efficacy; Polymorphism
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Intervention Model Description: 100 hepatocellular carcinoma patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sorafenib group (Experimental): 100 patients diagnosed with HCC for whom Sorafenib therapy is prescribed (400 mg twice daily) or (200mg twice daily), will be recruited from Mansoura University Hospital, Mansoura, Egypt.
  Interventions: Drug: Sorafenib Tablets

INTERVENTIONS:
Drug: Sorafenib Tablets — Sorafenib Tablets (200 -400 mg) twice daily
  Other Names: Nexavar

SUMMARY:
This study aims to determine the predictive effect of ATG10 and IL6 genetic polymorphisms in safety and efficacy of sorafenib used for the treatment of Egyptian HCC patients. Moreover, this study will determine the association between genetic polymorphisms of ATG10 and IL6 with HCC severity.

DETAILED DESCRIPTION:
A prospective pharmcogentic study for Egyptian HCC patients treating with oral sorafenib.

1. Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University.
2. 100 patients diagnosed with HCC for whom Sorafenib therapy is prescribed (400 mg twice daily) or (200mg twice daily),. will be recruited from Mansoura University Hospital, Mansoura, Egypt.
3. At baseline and follow up visits after Sorafenib, all patients will be assessed for complete blood count (CBC), kidney function, liver function, liver enzymes, alpha fetoprotein (AFP) and viral markers. Moreover, triphasic pelviabdominal CT will be performed .
4. Blood samples will be collected for ATG10 AND IL6 genotyping.
5. Genetic polymorphisms of ATG10 AND IL6 will be detected by real time polymerase chain reaction (RT-PCR).

   * Five mls of whole blood will be collected
   * Extraction of genomic DNA from blood samples by DNA extraction kit.
   * DNA qualification will be performed by Nano drop.
   * Genotyping will be done by allelic discrimination using Taqman assays specific for each polymorphism.
   * Assays will be done according to manufacturer protocol using real time PCR machine.
6. Appropriate statistical tests will be conducted to evaluate the significance of the results.
7. Results, conclusion, discussion and recommendations will be given. Ethical Issue

   * Informed consent will be signed by all eligible patients before enrolling in the study.
   * All patients' data will be confidential.

Efficacy and Safety outcomes:

1. Target lesions response will be measured according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) Complete response, Partial response, Progressive disease and Stable disease.
2. The appropriate dose of sorafenib will be determined individually based on the patient tolerability.
3. Follow up will be performed for detection of tumor size using triphasic CT scan as a measure of efficacy. Moreover, all patients will be reevaluated for CBC,AFP, liver and kidney functions, in the follow up visit, to detect incidence of any adverse effects.
4. Patients will be asked for any side effects such as (diarrhea, anorexia, nausea, vomiting).
5. Patients will be followed for progression-free survival after receiving soarfenib.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosed HCC patient.
2. Child-pugh class A.
3. Performance status 1-2 (ECOG scale)
4. Laboratory investigation : Hemoglobin ≥8.5 mg\dl, INR ≤2.3 ,Albumin≥2.8g\dl, ALT and AST ≤ 3 times the ULN
5. Age ≥20 years.

Exclusion Criteria:

1. Patients refused to sign the written consent.
2. Age > 75 years.
3. Renal failure requiring hemo- or peritoneal dialysis
4. History of cardiac disease
5. Active clinically serious infections
6. Known history of human immunodeficiency virus (HIV) infection
7. Pregnant female
8. Child-pugh class B and C.
9. Performance status 3 or 4.
10. Patient who are indicated for surgical resection or liver transplant (MDT).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
ATG10 genotyping | 6 months
  Gene polymorphism
IL6 genotyping | 6 months
  Gene polymorphism
Safety Outcomes | 6 months
  Incidence of side effects such as (diarrhea, anorexia, nausea, vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass. Prof., Study Chair — Damanhour University; Noha El bassiouny, Lecturer, Study Director — Damanhour University
Locations (1):
- Mansoura University Hospital, Al Mansurah, El-Dakahelia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Sheshtawy AM, Werida RH, Bahgat MH, El-Etreby S, El-Bassiouny NA. Pharmacogenomic insights: IL-23R and ATG-10 polymorphisms in Sorafenib response for hepatocellular carcinoma. Clin Exp Med. 2025 Feb 8;25(1):51. doi: 10.1007/s10238-025-01576-4. PMID 39921803